CLINICAL TRIAL: NCT01995266
Title: A Phase 3, Open-Label Study With Daclatasvir And Asunaprevir (DUAL) for Subjects With Genotype 1b Chronic Hepatitis C (HCV) Infection Who Are Intolerant or Ineligible to Interferon Alfa Therapies With or Without Ribavirin
Brief Title: Phase III China GT 1b Interferon (IFN) Intolerant Prev Exclude Dual
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AI447-036
Record Dates: First submitted 2013-11-21; First posted 2013-11-26 (Estimated); Results first posted 2019-07-11 (Actual); Last update posted 2020-08-11 (Actual); Status verified 2020-08

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C | interventions — asunaprevir; daclatasvir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Asunaprevir + Daclatasvir (Experimental): Asunaprevir 100mg soft capsule by mouth twice daily for 24 weeks and
  Daclatasvir 60mg tablet by mouth once daily for 24 weeks
  Interventions: Drug: Asunaprevir; Drug: Daclatasvir

INTERVENTIONS:
Drug: Asunaprevir
  Other Names: BMS-650032
Drug: Daclatasvir
  Other Names: BMS-790052

SUMMARY:
Patients with chronic hepatitis genotype 1b, who are intolerant or ineligible to Interferon alfa therapy with or without Ribavirin, will be treated for 24 weeks with Daclatasvir (DCV) Dual regimen (= Daclatasvir + Asunaprevir) and followed for an additional 24 weeks post-treatment in order to determine the safety and efficacy of the DCV DUAL regimen

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Males and females, ≥ 18 years of age
* Subjects chronically infected with HCV Genotype (GT)-1b only as documented by positive HCV RNA and anti-HCV antibody at screening and either:

  1. Positive anti-HCV antibody, HCV RNA or positive HCV genotype test at least 6 months prior to screening

     or
  2. Liver biopsy consistent with chronic HCV infection (evidence of fibrosis and/or inflammation)
* Subjects who are intolerant to previous therapy with Interferon Alfa (IFNα) either with or without Ribavirin (RBV) (I±R)(independent of previous response to therapy) or ineligible for I±R and who meet one of the criteria below:

  1. Anemia: the I±R intolerants are subjects who were previously treated with IFNα/RBV therapy and had a decline in hemoglobin to < 8.5 g/dL during therapy (documented); the I±R ineligibles are subjects who have a screening hemoglobin < 10.0 g/dL and ≥ 8.5 g/dL

     OR
  2. Neutropenia: the I±R intolerants are subjects who were previously treated with IFNα/RBV therapy and had a decline in absolute neutrophil count (ANC) to < 0.5 x 10(9) during therapy (documented); the I±R ineligibles are subjects who have a screening ANC < 1.5 x 10(9) cells/L and ≥ 0.5 x 10(9) cells/L

     OR
  3. Thrombocytopenia: the I±R intolerants are subjects who were previously treated with IFNα/RBV therapy and had a decline in platelet counts < 25,000 cells/mm3 during therapy (documented); the I±R ineligibles are subjects who have a screening platelet count of < 90 x 10(9) cells/L and ≥ 50 x 10(9) cells/L
* HCV RNA ≥ 10,000 IU/mL
* Seronegative for Human Immunodeficiency Virus (HIV) and hepatitis B surface antigen (HBsAg)
* Body Mass Index (BMI) of 18 to 35 kg/m2, inclusive. BMI = weight (kg)/ [height(m)]2 at screening
* Subjects with compensated cirrhosis are permitted (compensated cirrhotics are capped at approximately 40%). If a subject does not have cirrhosis, a liver biopsy within three years prior to enrollment is required to demonstrate the absence of cirrhosis. If cirrhosis is present, any prior liver biopsy is sufficient. For countries where liver biopsy is not required prior to treatment and where noninvasive imaging tests (Fibroscan® ultrasound) are approved for staging of liver disease, non-invasive imaging test results may be used to assess the extent of liver disease

Exclusion Criteria:

* Prior treatment with HCV direct acting antiviral (DAA)
* Evidence of a medical condition contributing to chronic liver disease other than HCV
* Evidence of decompensated liver disease including, but not limited to, a history or presence of ascites, bleeding varices, or hepatic encephalopathy
* Diagnosed or suspected hepatocellular carcinoma or other malignancies
* Uncontrolled diabetes or hypertension
* History of moderate to severe depression. Well-controlled mild depression is allowed
* Total bilirubin ≥ 34 µmol/L (or ≥ 2 mg/dL) unless subject has a documented history of Gilbert's disease
* Confirmed alanine aminotransferase (ALT) ≥ 5 x upper limit of normal (ULN)
* Confirmed albumin < 3.5 g/dL (35 g/L)
* Alpha-fetoprotein (AFP) > 100 ng/mL OR ≥ 50 and ≤ 100 ng/mL requires a liver ultrasound and subjects with findings suspicious of hepatocellular carcinoma (HCC) are excluded
* Confirmed hemoglobin < 8.5 g/dL
* Confirmed ANC < 0.5 x 10(9) cells/L
* Confirmed platelet count < 50,000 cells/mm3

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 218 (Actual)
Dates: Start 2014-02-28 (Actual); Primary Completion 2015-07-31 (Actual); Study Completion 2015-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (27):
- China (16):
  - Local Institution, Beijing, Beijing Municipality
  - Local Institution, Beijing, Guangdong
  - Local Institution, Chongqing, Guangdong
  - Local Institution, Guangzhou, Guangdong
  - Local Institution, Wuhan, Hubei
  - Local Institution, Changsha, Hunan
  - Local Institution, Nanjing, Jiangsu
  - Local Institution, Changchun, Jilin
  - Local Institution, Shenyang, Liaoning
  - Local Institution, Xi'an, Shan3xi
  - Local Institution, Shanghai, Shanghai Municipality
  - Local Institution, Beijing, Shanxi
  - Local Institution, Shanghai, Shanxi
  - Local Institution, Tianjin, Tianjin Municipality
  - Local Institution, Beijing
  - Local Institution, Chongqing
- South Korea (7):
  - Local Institution, Seoul, Beijing
  - Local Institution, Busan, Guangdong
  - Local Institution, Seoul, Guangdong
  - Local Institution, Daegu, Hunan
  - Local Institution, Busan
  - Local Institution, Daegu
  - Local Institution, Seoul
- Taiwan (4):
  - Local Institution, Kaohsiung City, Guangdong
  - Local Institution, Tainan, Guangdong
  - Local Institution, Kaohsiung City
  - Local Institution, Tainan

REFERENCES:
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 218 participants enrolled, 159 were treated. Of the 59 who were not treated, 55 did not meet study criteria and 4 withdrew consent to participate.
Groups:
- All Subjects: Oral dose of daclatasvir (DCV) 60 mg once daily (QD) and asunaprevir (ASV) 100 mg twice daily (BID) was administered for 24 weeks. Thereafter, participants entered a follow-up period of 24 weeks after completion of study treatment or upon early discontinuation of treatment.
Period: Overall Study
Arm/Group | All Subjects
Started | 159
Completed | 150
Not Completed | 9
Not completed — Death | 1
Not completed — Lack of Efficacy | 6
Not completed — Adverse Event | 2

BASELINE CHARACTERISTICS:
Population: All treated participants.
Arm/Group | All Subjects
Number analyzed (Participants) | 159
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.6 (12.30)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 104
  Male | 55
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 159
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Virologic Response (SVR) at Post-Treatment Follow-up Week 24 (SVR24)
Description: SVR was defined as Hepatitis C Virus ribonucleic acid (HCV RNA) < lower limit of quantitation (LLOQ) target detected (TD) or not detected (TND) at post-treatment follow-up Week 24.
Time Frame: 24 Weeks after treatment discontinuation (Follow-up Week 24)
Population: All treated and evaluable participants.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | All Subjects
Number analyzed (Participants) | 159
Percentage of participants | 91.2 [85.7 to 95.1]

2. Secondary Outcome: Percentage of Participants With Sustained Virologic Response (SVR) at Post-Treatment Follow-up Week 12 (SVR12)
Description: SVR12 was defined as HCV RNA < LLOQ target detected or not detected at post-treatment follow-up Week 12. For SVR12, missing HCV RNA data at follow-up Week 12 was imputed using the Next Value Carried Backwards (NVCB) approach.
Time Frame: 12 Weeks after treatment discontinuation (Follow-up Week 12)
Population: All treated and evaluable participants.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | All Subjects
Number analyzed (Participants) | 159
Percentage of participants | 91.2 [85.7 to 95.1]

3. Secondary Outcome: Number of Participants With Adverse Events (AEs), Serious AEs (SAEs), Death, and AEs Leading to Discontinuation
Description: An AE is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An AE can therefore be any unfavorable and unintended sign (example, a clinically significant abnormal laboratory finding), symptom, or disease temporally associated with the use of a drug, whether or not it is considered related to the drug. An SAE is an AE resulting in any of the following outcomes or deemed significant for any other reason: death, initial or prolonged inpatient hospitalization, life-threatening experience (immediate risk of dying), persistent or significant disability/incapacity, or a congenital anomaly, or a medically important event.
Time Frame: 7 days after treatment discontinuation
Population: All treated and evaluable participants.
Measure: Count of Participants; unit: Participants
Arm/Group | All Subjects
Number analyzed (Participants) | 159
Participants
  Death | 1
  SAEs | 5
  AEs | 118
  AEs leading to discontinuation | 2

4. Secondary Outcome: Percentage of Participants With SVR24 by the rs12979860 Single Nucleotide Polymorphisms (SNP) in the IL 28B Gene at Post-Treatment Follow-up Week 24
Description: Participants categorized into three genotypes based on SNPs in the IL28B gene were assessed for SVR24, defined as response in which hepatitis C virus RNA levels below lower limit of quantitation or below target detected or target not detected at follow-up Week 24.
Time Frame: 24 Weeks after treatment discontinuation (Follow-up Week 24)
Population: All evaluable participants of each Genotype who received treatment
Measure: Number; unit: Percentage of participants
Arm/Group | All Subjects
Number analyzed (Participants) | 159
Percentage of participants
  CC Genotype: number analyzed (Participants) | 95
  CC Genotype | 89.5
  CT Genotype: number analyzed (Participants) | 57
  CT Genotype | 93.0
  TT Genotype: number analyzed (Participants) | 7
  TT Genotype | 100

5. Secondary Outcome: Percentage of Participants With HCV RNA< LLOQ Target Not Detected at the End of Treatment (Week 24)
Description: Blood was drawn from each participant to assess HCV RNA plasma levels using the Roche COBAS® Taqman quantitative RT-PCR assay, v2.0. The lower and upper limits of quantitation (LOQs) of the assay for HCV GT-1 were 25 IU/mL and 3.91 X10^8 IU/mL, respectively; the limit of detection was ~ 10 IU/mL
Time Frame: Week 24 (End-of Treatment)
Population: All treated and evaluable participants.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | All Subjects
Number analyzed (Participants) | 159
Percentage of participants | 92.5 [87.2 to 96.0]

6. Secondary Outcome: Number of Participants With Rapid Virologic Response (RVR)
Description: RVR was defined as HCV RNA < LLOQ, target not detected at treatment Week 4.
Time Frame: Treatment Week 4
Population: All treated and evaluable participants.
Measure: Count of Participants; unit: Participants
Arm/Group | All Subjects
Number analyzed (Participants) | 159
Participants | 136

7. Secondary Outcome: Percentage of Participants With Complete Early Virologic Response (cEVR)
Description: cEVR was defined as HCV RNA < LLOQ, target not detected at treatment Week 12.
Time Frame: Treatment Week 12
Population: All treated and evaluable participants.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | All Subjects
Number analyzed (Participants) | 159
Percentage of participants | 96.2 [92.0 to 98.6]

8. Secondary Outcome: Number of Participants With Extended Rapid Virologic Response (eRVR)
Description: eRVR was defined as HCV RNA < LLOQ, target not detected at treatment Weeks 4 and 12.
Time Frame: Treatment Week 4 and Week 12
Population: All treated and evaluable participants.
Measure: Count of Participants; unit: Participants
Arm/Group | All Subjects
Number analyzed (Participants) | 159
Participants | 134

9. Secondary Outcome: Number of Participants With HCV RNA < LLOQ Target Detected or Not Detected at the End of Treatment (Week 24)
Description: Antiviral efficacy is measured by the number of participants with HCV RNA< LLOQ (lower limit of quantification), TD (target detected) or TND (target not detected) at End of Treatment (Week 24)
Time Frame: Week 24 (End-of Treatment)
Population: All treated and evaluable participants.
Measure: Count of Participants; unit: Participants
Arm/Group | All Subjects
Number analyzed (Participants) | 159
Participants | 149

10. Secondary Outcome: Number of Participants With Virologic Response (VR) at Treatment Week 4 and 12
Description: VR was defined as HCV RNA < LLOQ, target detected or not detected at specific time points (Week 4 and Week 12)
Time Frame: Treatment Week 4 and 12
Population: All treated and evaluable participants.
Measure: Count of Participants; unit: Participants
Arm/Group | All Subjects
Number analyzed (Participants) | 159
Participants | 151

ADVERSE EVENTS:
Time Frame: Up to 24 weeks within 30 days of discontinuation of dosing
Description: Analysis was performed on all treated participants.
Arm/Group | All Subjects
All-Cause Mortality (participants affected / at risk) | 1/159
Serious Adverse Events (participants affected / at risk) | 5/159
Other Adverse Events (participants affected / at risk) | 66/159
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Subjects (N=159)
Adam-Stokes Syndrome (Cardiac disorders) | 1
Asteriosclerosis Coronary Artery (Cardiac disorders) | 1
Coronary Artery Disease (Cardiac disorders) | 1
Sudden Hearing Loss (Ear and labyrinth disorders) | 1
Pneumonia (Infections and infestations) | 1
Femoral Neck Fracture (Injury, poisoning and procedural complications) | 1
Hepatocellular Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Arrhythmia (Cardiac disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | All Subjects (N=159)
Platelet Count Decreased (Investigations) | 14
Alanine Aminotransferase Increased (Investigations) | 11
Neutrophil Count Decreased (Investigations) | 11
Monocyte Count Decreased (Investigations) | 10
White Blood Cell Count Decreased (Investigations) | 10
Aspartate Aminotransferase Increased (Investigations) | 8
Upper Respiratory Tract Infection (Infections and infestations) | 13
Thrombocytopenia (Blood and lymphatic system disorders) | 10
Pruritus (Skin and subcutaneous tissue disorders) | 9
Diarrhoea (Gastrointestinal disorders) | 8
Hyperuricaemia (Metabolism and nutrition disorders) | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submitting for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.